CLINICAL TRIAL: NCT07239635
Title: Effect of Perch Essence on Cognitive Function Status in Subjects With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202401063
Record Dates: First submitted 2025-11-13; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Control group were asked to maintain their dietary habit, lifestyle, and used of medication, and were provided 60 mL/packet, twice daily for 24 weeks of fish stock with the same appearance, flavor, and color similar to perch essence as placebo.
  Interventions: Dietary Supplement: Fish stock
- Perch essence (Experimental): Treatment group were asked to maintain their dietary habit, lifestyle, and used of medication, and were provided 60 mL/packet, twice daily for 24 weeks of perch essence.
  Interventions: Dietary Supplement: Perch essence

INTERVENTIONS:
Dietary Supplement: Perch essence — 60mL/packet of perch essence, twice daily for 24 weeks
  Arms: Perch essence
Dietary Supplement: Fish stock — 60mL/packet of fish stock, twice daily for 24 weeks, with the same appearance, flavor, and color compared to perch essence
  Arms: Placebo

SUMMARY:
With global population aging, cognitive impairment and dementia have become major public health issues worldwide. According to the 2019 World Alzheimer Report by the Alzheimer's Disease International, there are more than 50 million people living with dementia globally, and this number is projected to rise to 152 million by 2050, with one new case occurring every three seconds. Our research is to investigate the intervention effects of perch essence on cognitive function in mild-cognitive impairment patients.

1. Study population: 54 MCI patients were recruited and the inclusion criteria are: (1) aged ≥ 45, (2) diagnosed with mild cognitive impairment by clinical dementia rating (CDR) with a scoring of 0.5, and (3) have the ability to communicate, reading and writing. The exclusion criteria are: (1) diagnosed with dementia, (2) diagnosed with terminal diseases or severe psychological symptoms (lifespan ≤ 2 years, cancer, severe stroke, heart disease, liver cirrhosis, ESRD, severe depression, etc.), (3) Severe blindness, hearing impairment, or communication disability, (4) Branched-chain organic aciduria (e.g., maple syrup urine disease), (5) Individuals who do not consume fish or are allergic to fish products 2. Study design: A two-arm single-blind randomized controlled clinical trial will be performed for 24 weeks and the subjects will be divided in to 2 groups: (1) control group, (2) treatment group. S The treatment group were asked to consume 60mL/packet of perch essence, twice daily for 24 weeks, whereas the control group were provided with the same appearance, flavor, and color of fish stock. Participants were asked to maintain their dietary habit, lifestyle, and used of medication.

3. Outcome assessment:

1. Anthropometry data: height, weight, body mass index
2. Blood biochemistry:

   A. Nutritional status: albumin, total protein, Vitamin B12, folate, magnesium B. Glycemic profiles: fasting blood glucose C. Lipid profiles: total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), triglycerides (TG).

   D. Complete blood counts: white blood cells (WBC), red blood cells (RBC), hemoglobin (HB), platelet count (PLT), hematocrit (HCT), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC).

   E. Brain derived neurotrophic factor (BDNF), malondialdehyde (MDA)
3. Urine test Urine color, appearance, specific gravity, pH, glucose, creatinine
4. Cognitive function: Montreal cognitive assessment (MoCA), Cognitive abilities screening instruments (CASI)
5. Nutrition status Mini-nutritional assessments (MNA), 3-day dietary recall The purpose of the study investigated the intervention of perch essence supplement on cognitive function and its correlation with nutritional status in MCI patients.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 45
* diagnosed with mild cognitive impairment by clinical dementia rating (CDR) with a scoring of 0.5
* have the ability to communicate, reading and writing

Exclusion Criteria:

* diagnosed with dementia
* diagnosed with terminal diseases or severe psychological symptoms (lifespan ≤ 2 years, cancer, severe stroke, heart disease, liver cirrhosis, ESRD, severe depression, etc.)
* Severe blindness, hearing impairment, or communication disability
* Branched-chain organic aciduria (e.g., maple syrup urine disease)
* Individuals who do not consume fish or are allergic to fish products

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Cognitive Abilities Screening Instrument (CASI) | Week 0, 12, and 24
  Cognitive assessments, ranges from 0 to 100, with higher scores indicating better cognitive function, lower than 74 may indicate cognitive impairment, and scores are also affected by age and education level.
Montreal Cognitive Assessment | Week 0, 12, and 24
  Cognitive assessments, 30 score as full, scoring ≥26 considered as normal, below 26 may indicate impairment, with a score of 18-25 suggesting mild impairment, 10-17 moderate impairment, and below 10 indicating severe impairment.

SECONDARY OUTCOMES:
Anthropometric data | Week 0, 12, and 24
  Weight and height will be combined to calculate BMI (kg/m2)
Blood biochemistry: Nutritional status | Week 0, 12, and 24
  Albumin, total protein, Vitamin B12, folate, magnesium
Blood biochemistry: Glycemic profiles | Week 0, 12, and 24
  fasting blood glucose
Blood biochemistry: Lipid profiles | Week 0, 12, and 24
  total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), triglycerides (TG)
Blood biochemistry: Complete blood counts | Week 0, 12, and 24
  white blood cells (WBC), red blood cells (RBC), hemoglobin (HB), platelet count (PLT), hematocrit (HCT), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC)
Blood biochemistry: BDNF and oxidative stress | Week 0, 12, and 24
  Brain derived neurotrophic factor (BDNF), malondialdehyde (MDA)
Nutrition status | Week 0, 24
  Mini-nutritional assessments (MNA): Maximum scores are at 30; scores ≥ 24: not in malnutrition risk; 17-23.5: risk in malnutrition, <17: malnutrition.
  3-day dietary recall

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nutrition and Health Sciences, Taipei, Xinyi, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided